CLINICAL TRIAL: NCT04896840
Title: The Effect of Motor Learning Based Tele-rehabilitation on Quality of Life in Children With Cerebral Palsy During the Covid-19 Epidemic Process
Brief Title: Tele-rehabilitation in Children With Cerebral Palsy in the Covid-19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Engin Ramazanoglu, Researcher, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/1422
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy; Telerehabilitation; Motor Learning
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Telerehabilitation and motor learning principles will be applied.
  Interventions: Other: Telerehabilitation İntervention, Motor learning
- Control Group (Experimental): Motor learning principles will be applied in the clinic.
  Interventions: Other: Telerehabilitation İntervention, Motor learning

INTERVENTIONS:
Other: Telerehabilitation İntervention, Motor learning — Telerehabilitation İntervention:
  Training videos will be sent to the families of the children in the tele-rehabilitation group before starting to work. With the training videos, it is aimed to teach the exercises to be done to the families. Treatment will be applied by their families for 8 weeks, 2 days a week, 40 minutes a day. Physiotherapist will attend the sessions by video conference method. Video conference calls will be made by phone over the WhatsApp application.
  Motor learning:
  The first 10 minutes will start with active stretching Functional lying in a sitting position, Functional lying with feet together in a standing position. rolling the pilates ball on the wall, walking on its side. Going up and down stairs at different heights. Walking across different surfaces and obstacles. Getting up from chairs of different heights, sitting and extending the object taken from the ground. Functional exercises suitable for the child's level.

SUMMARY:
The investigators study aimed to observe the effect of motor learning-based tele-rehabilitation on quality of life in children with cerebral palsy during the Covid-19 pandemic.

DETAILED DESCRIPTION:
Cerebral palsy; It is defined as a permanent, non-progressive disorder that occurs as a result of the effects of the developing fetal or infant brain for different reasons in prenatal, perinatal or postnatal periods. Children with cerebral palsy experience fundamental limitations in the postural control of static and dynamic tasks such as sitting, standing, and walking. However, children with cerebral palsy need rehabilitation. The COVID-19 pandemic prevents effective provision of rehabilitation services for children with cerebral palsy. However; Lack of access to rehabilitation services in individuals with cerebral palsy during the COVID-19 pandemic has increased the need for alternative and complementary methods. During the Covid-19 pandemic process, the tele-rehabilitation process will be able to achieve functional and social participation in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children with spastic cerebral palsy, ages 3-16
* To be at 1-2-3 levels according to GMFCS
* The tele-rehabilitation group is not receiving treatment in any center.
* Voluntary participation in the study with the consent of the parents

Exclusion Criteria:

* Application of muscle tone reduction 6 months before the start of the study (eg botulin toxin, baclofen pump therapy) or those undergoing orthopedic surgery.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Estimated)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory | 8 weeks
  The 35-item PedsQL consists of seven subscales: Daily Activities, School Activities, Movement and Balance, Pain, Fatigue, Eating Activities, Speaking and Communication. The scale consists of a child self-report and a parent report. The scale questions the degree of problems the children have experienced in the last month. Item scores are converted linearly backwards on a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so higher scores indicate better health-related quality of Life.Subscale scores are calculated by dividing the total score of the items answered by the number of items answered. There is no scale total score, subscales have calculated mean scores. The higher the average score for an area (subscale) indicates that there are fewer problems in that area and the higher the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The information of the patients participating in the study will be kept confidential.

REFERENCES:
- [Background] Bar-Haim S, Harries N, Nammourah I, Oraibi S, Malhees W, Loeppky J, Perkins NJ, Belokopytov M, Kaplanski J, Lahat E; MERC project. Effectiveness of motor learning coaching in children with cerebral palsy: a randomized controlled trial. Clin Rehabil. 2010 Nov;24(11):1009-20. doi: 10.1177/0269215510371428. Epub 2010 Jun 24. PMID 20576667
- [Background] Dunn AM, Patel KP. Integration of geriatric with general medical services. Lancet. 1983 Nov 12;2(8359):1139. doi: 10.1016/s0140-6736(83)90650-5. No abstract available. PMID 6138665
- [Background] Meijer HA, Graafland M, Goslings JC, Schijven MP. Systematic Review on the Effects of Serious Games and Wearable Technology Used in Rehabilitation of Patients With Traumatic Bone and Soft Tissue Injuries. Arch Phys Med Rehabil. 2018 Sep;99(9):1890-1899. doi: 10.1016/j.apmr.2017.10.018. Epub 2017 Nov 11. PMID 29138050
- [Background] Pastora-Bernal JM, Martin-Valero R, Baron-Lopez FJ, Estebanez-Perez MJ. Evidence of Benefit of Telerehabitation After Orthopedic Surgery: A Systematic Review. J Med Internet Res. 2017 Apr 28;19(4):e142. doi: 10.2196/jmir.6836. PMID 28455277
- [Background] Woollacott MH, Shumway-Cook A. Postural dysfunction during standing and walking in children with cerebral palsy: what are the underlying problems and what new therapies might improve balance? Neural Plast. 2005;12(2-3):211-9; discussion 263-72. doi: 10.1155/NP.2005.211. PMID 16097489